CLINICAL TRIAL: NCT04431245
Title: Stopping Antiviral Treatment and Subsequent Flare in Chronic Hepatitis B Infection: Immunological and Virological Profiling
Brief Title: Stopping Antiviral Treatment in Chronic Hepatitis B
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yuen Man Fung, Chair Professor, The University of Hong Kong
Other Study IDs: HKUUW20-425
Record Dates: First submitted 2020-05-31; First posted 2020-06-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Hepatitis b
Keywords: functional cure; antiviral therapy; nucleoside analogue
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Nucleosides

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stop antiviral: HBeAg-negative non-cirrhotic CHB patients on long-term NA ≥3 years will be identified. Only those who have undetectable serum HBV DNA by the conventional assay (Cobas Taqman, Roche Diagnostics, Branchburg, NJ) which has a lower limit of detection (LLOD) of 10 IU/mL will be recruited. CHB patients were treated with potent oral NA (i.e. tenofovir or entecavir). All recruited patients will have written informed consent for participation of study. Patients with HCC, cirrhosis, history of liver transplantation, or on immunosuppressants, will be excluded.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Study subjects will stop the antiviral therapy. Patients will be closely monitored every 6-8 weeks for virological flare and/or biochemical flare.
  Other Names: oral nucleoside analogue

SUMMARY:
Chronic hepatitis B (CHB) infection affected 292 million individuals in the world, translating to about 3.9% of global prevalence. Up to 40% of patients with CHB will develop liver-related complications. Many patients require long-term oral antiviral therapy since off-treatment sustained virological control can only be achieved in a minority of patients. It is uncommon for patients taking long-term antivirals to be able to stop the treatment if favorable factors are not present. Those include low viral load, long enough duration of treatment, and absence of cirrhosis. Some studies have found that inducing a mild flare is beneficial for achieving functional cure in chronic hepatitis B infection. There is lack of data in the immunological and virological profile in patients who stop their long-term antiviral therapy, and in those who developed flare after treatment cessation.

DETAILED DESCRIPTION:
Chronic hepatitis B infection (CHB) affected 292 million individuals in the world in 2016 according to the Polaris Observatory estimation, translating to about 3.9% global prevalence. Up to 40% of patients with CHB will develop liver-related complications and there were 890,000 deaths from these complications in 2015. Current antiviral therapy is aimed to achieve effective viral suppression, biochemical remission, histological improvement, and risk reductions in liver-related complications including cirrhosis and liver cancer. Many patients require long-term oral nucleos(t)ide analogues (NA) since off-treatment sustained virological control can only be achieved in a minority of patients. For HBeAg-negative CHB patients, variable rates of durable virological response were observed after cessation of NA. Only a small proportion of HBeAg-negative Asian patients (<10%) can successfully stop NA without virological breakthrough, compared to more than 60% of Caucasian patients maintaining a durable virologic response and even HBsAg seroclearance in up to 30%. Therefore, current guidelines in general recommend indefinite duration of NA therapy in HBeAg-negative patients, unless guaranteed close monitoring could be provided after cessation of NA in suitable subjects. Favourable factors predictive of partial cure include lower baseline HBV DNA, lower HBsAg titre or hepatitis B core-related antigen at NA cessation and longer duration of consolidation therapy in HBeAg-negative patients. There is lack of data in the immunological and virological profile in patients who stop their long-term NA, and in those who developed post-NA cessation flare.

The investigators aim to study the virological and immunological profile in patients who stopped long-term NA therapy, with or without post-NA cessation flare. In addition, the investigators would like to investigate the effect of mild flare after monitored NA-cessation on subsequent virological activity and HBsAg seroclearance.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg-negative
* non-cirrhotic
* on long-term NA ≥3 years (entecavir or tenofovir)
* undetectable serum HBV DNA

Exclusion Criteria:

* HCC, cirrhosis, history of liver transplantation, or on immunosuppressants,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBeAg-negative non-cirrhotic CHB patients on long-term NA ≥3 years will be identified. Only those who have undetectable serum HBV DNA by the conventional assay (Cobas Taqman, Roche Diagnostics, Branchburg, NJ) which has a lower limit of detection (LLOD) of 10 IU/mL will be recruited. CHB patients were treated with potent oral NA (i.e. tenofovir or entecavir). All recruited patients will have written informed consent for participation of study. Patients with HCC, cirrhosis, history of liver transplantation, or on immunosuppressants, will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The immunological profile in CHB patients who stopped antiviral therapy | 24 months
  The investigators will perform analysis for the immunological aspects for these patients
The virological profile in CHB patients who stopped antiviral therapy | 24 months
  The investigators will perform analysis for the virological aspects for these patients

CONTACTS AND LOCATIONS:
Overall Officials: Man-Fung Yuen, DSc, MD, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Man Fung Yuen, Hong Kong, Please Select One ..., Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant's personal identification data will be only accessed by the PI and study team.